CLINICAL TRIAL: NCT03721081
Title: Preemptive Local Anesthetic Infiltration Reduces Opioid Requirements Without Attenuation of the Intraoperative Evoked Stapedial Reflex Thresholds in Pediatric Cochlear Implant Surgery
Brief Title: Local Anesthesia for Pediatric Cochlear Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: Bahteem Specialized Hospital (Other)
Responsible Party: Sponsor-Investigator, Wahba bakhet, Lecturer, Ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WBAKHET-LA
Record Dates: First submitted 2018-10-17; First posted 2018-10-26 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Na Cl 0.9%/Epi 1:200000 (Placebo Comparator): Subcutaneous infiltration of Na Cl 0.9%/Epi 1:200000
  Interventions: Other: Na Cl 0.9%/Epi 1:200000
- Lidocaine 1%/Epi 1:200000 (Active Comparator): Subcutaneous infiltration of Lidocaine 1%/Epi 1:200000
  Interventions: Drug: Lidocaine 1%/Epi 1:200000

INTERVENTIONS:
Drug: Lidocaine 1%/Epi 1:200000 — Five minutes before skin incision, subcutaneous infiltration of 0.5 ml/kg of Lidocaine 1%/Epi 1:200000 Inj along a 3 cm extended endaural incision with a 23 G hypodermic needle administered was performed by the surgeon, who was blinded to the applied drug solution.
  Other Names: Xylocaine 1%/Epi 1:200000
  Arms: Lidocaine 1%/Epi 1:200000
Other: Na Cl 0.9%/Epi 1:200000 — Five minutes before skin incision, subcutaneous infiltration of 0.5 ml/kg of Na CI 0.9%/Epi 1:200000 inj along a 3 cm extended endaural incision with a 23 G hypodermic needle administered was performed by the surgeon, who was blinded to the applied drug solution.
  Arms: Na Cl 0.9%/Epi 1:200000

SUMMARY:
Propofol with remifentanil provides good operative conditions for pediatric cochlear implant (CI); however, large doses of remifentanil usually result in postoperative hyperalgesia and increase postoperative pain. Local anesthesia (LA) is commonly used as an adjunct to general anesthesia in children; however, otologists are usually reluctant in the use of LA as it can cause abolishment of the electrical stapedial reflex threshold (ESRT).

DETAILED DESCRIPTION:
Seventy children (1-6 years) undergoing CI were recruited. Children were divided into two groups. The LA group received subcutaneous infiltration of 0.5 ml/kg lidocaine 1% in adrenaline 1:200,000 and the CT group received 0.5 ml/kg of Na CI 0.9% in adrenaline 1:200,000. The primary outcome was number of patients requiring rescue analgesia (tramadol) during the first 24-h postoperative. Secondary outcomes were haemodynamic variables, the ESRT, intraoperative anesthetic requirements, time to LMA removal, time to total recovery, pain scores, time to first rescue analgesia and incidence of vomiting.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status,
* age between 1 and 6 year,

Exclusion Criteria:

* known allergy to local anesthetics,
* predicted operative difficulty (i.e. syndromic hearing loss, congenital cochlear abnormalities or cochlear ossification.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
number of patients requiring rescue opioid analgesia (Tramal) | During the length of hospital stay post surgery (on average 24 hours)
  Post-operative Pain assessed by the pediatric observational Faces, Legs, Activity, Cry Consolability (FLACC) score with its 0 to 10 score range: (0 (no pain) to 10 ( Severe pain)

SECONDARY OUTCOMES:
The operative time | Intraoperative
  Minutes
The anesthesia time. | Intraoperative
  Minutes
Heart rate | Intraoperative
  beats per minute
mean arterial blood pressure | Intraoperative
  mm Hg
ESRT responses | Intraoperative
  The surgeon assessed ESRT response at the basal, middle, and apical areas of the electrode array by visual monitoring of the stapedius muscle using direct microscopic examination
Anesthetic consumption | Intraoperative
  propofol and remifentanil requirement after the bolus

CONTACTS AND LOCATIONS:
Overall Officials: wahba Z Bakhet, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided